CLINICAL TRIAL: NCT02727777
Title: Phase II Study of TAK228 in Relapsed Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0501; NCI-2016-00671 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-03-25; First posted 2016-04-05 (Estimated); Results first posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Lymphoma
Keywords: Lymphoma; Relapsed Lymphoma; MLN0128; Blood sugar; Glucometer; TK228
MeSH Terms: conditions — Lymphoma | interventions — sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Aggressive Non-Hodgkin Lymphoma (NHL) - TAK228 (Experimental): Phase II - Aggressive NHL: Diffuse Large B Cell Lymphoma (DLBCL), Mantle Cell Lymphoma (MCL), Transformed Large Cell Lymphoma, and Follicular Lymphoma (FL) grade 3b Group
  Participants take TAK-228 1 time every day of a 28 day cycle.
  Treatment continues until progression of disease occurs, or a maximum of 12 months of treatment.
  Participant checks blood sugar every day before TAK-228 dose.
  Interventions: Drug: TAK228; Other: Blood Sugar Testing
- Indolent Non-Hodgkin Lymphoma (NHL) - TAK228 (Experimental): Phase II - Indolent NHL: Follicular Lymphoma (FL) grade 1-3a, Small Lymphocytic Lymphoma (SLL), Marginal Zone Lymphoma (MZL) Group
  Participants take TAK-228 1 time every day of a 28 day cycle.
  Treatment continues until progression of disease occurs, or a maximum of 12 months of treatment.
  Participant checks blood sugar every day before TAK-228 dose.
  Interventions: Drug: TAK228; Other: Blood Sugar Testing
- Hodgkin Lymphoma - TAK228 (Experimental): Phase II - Hodgkin Lymphoma Group
  Participants take TAK-228 1 time every day of a 28 day cycle.
  Treatment continues until progression of disease occurs, or a maximum of 12 months of treatment.
  Participant checks blood sugar every day before TAK-228 dose.
  Interventions: Drug: TAK228; Other: Blood Sugar Testing

INTERVENTIONS:
Drug: TAK228 — Starting dose of TAK228: 3 mg by mouth every day of a 28 day cycle.
  Other Names: MLN0128
Other: Blood Sugar Testing — Participant given a glucometer to check pre-dose blood sugar levels at home every day.

SUMMARY:
The goal of this clinical research study is to learn if TAK-228 can help to control relapsed lymphoma. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible for this study, you will begin taking capsules of TAK-228 in 28-day cycles. You will take the drug 1 time every day at about the same time. You should take the drug with about a cup (8 ounces) of water after eating a light meal. You should fast for 2 hours before and 1 hour after each dose.

If you vomit or have other digestive side effects that prevent you from taking a dose, that dose should be skipped. If you vomit up a dose, that dose should not be retaken. In both cases, wait until the next day to take another dose. In no case should you double or repeat a dose. You should record any vomiting in the dose diary the study staff provides you with.

Study Visits:

Within 3 days before you start taking TAK-228, blood (about 2 teaspoons) will be drawn for biomarker testing. Biomarkers are found in the blood/tissue and may be related to your reaction to the study drug.

On Day 1 of each cycle:

* You will have a physical exam.
* Blood (about 2-3 tablespoons) will be drawn for routine tests. You must fast for 4 hours before this blood draw. Some of these draws will be used for a diabetes test. If you can become pregnant, part of this sample will be used for a pregnancy test.
* Blood (about 2 teaspoons) will be drawn for biomarker testing (Cycles 1 and 2 only).
* You will have an EKG (within 3 days of each cycle after Cycle 1).

On Days 8 and 22 of Cycle 1, you will have a physical exam.

On Day 15 of Cycle 1:

* You will have a physical exam
* Blood (about 2-3 tablespoons) will be drawn for routine tests.

Within 5 days before Day 1 of Cycle 3, then every even-numbered cycle after that (Cycles 4, 6, 8, and so on), you will have CT scans, chest x-rays, and a bone marrow biopsy/aspiration to check the status of the disease.

If the study doctor thinks it is in your best interest, you will have PET/CT scans every 2 cycles to check the status of the disease.

Blood Sugar Testing:

You will be given a glucometer to check your pre-dose blood sugar levels at home every day. The study staff will teach you how to use the glucometer and what an abnormal reading looks like. You must tell the study staff right away if you have any abnormal readings. The frequency of in-home fasting glucose testing may be reduced to once weekly if the doctor thinks it is needed.

Length of Study:

You may continue to receive the study drug for up to 12 cycles. You will no longer be able to take the drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation in this study will be over after the follow-up phone calls have finished.

End-of-Treatment Visits:

About 1 week after you stop taking the study drug:

* You will have a physical exam
* Blood (about 2-3 tablespoons) will be drawn for routine tests and to test for diabetes. This will include a pregnancy test if you are able to become pregnant.
* You will have an EKG.

About 2 weeks after you stop taking the study drug, you will have CT scans and chest x-rays to check the status of the disease. If the study doctor thinks it is needed, you will also have a bone marrow biopsy/aspiration to check the status of the disease.

Within 2 weeks after you stop taking the study drug, blood (about 2 teaspoons) will be drawn for biomarker testing.

This is an investigational study. TAK-228 is not FDA approved or commercially available. It is currently being used for research purposes only. The study doctor can describe how the study drug is designed to work.

Up to 75 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Each patient must meet all of the following inclusion criteria to be enrolled in the study: 1. Male or female patients 18 years or older.
2. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
3. Female patients who: are postmenopausal for at least 1 year before the screening visit, OR are surgically sterile, OR if they are of childbearing potential, agree to practice 1 effective methods of contraception and one additional effective (barrier) method, at the same time, from the time of signing the informed consent through 90 days (or longer, as mandated bu local labeling [eg,USPI, SmPC, etc;]) after the last dose of study drug, or agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient (Periodic abstinence [e.g, calendar, ovulation, symptothermal, postovulation methods] and withdrawal,spermicides only, ad lactational amenorrhea are not acceptable methods of contraception.Female and male condoms should not be used together.
4. Male patients, even if surgically sterilized (ie, status post-vasectomy), who: agree to practice highly effective barrier contraception during the entire study treatment period and through 120 days after the last dose of study drug, or agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient (Periodic abstinence [e.g, calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal, spermicides only, ad lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together; Agree not to donate sperm during the course of this study or 120 days after receiving their last dose of study drug
5. Patients must have a diagnosis of prior treated diffuse large b-cell lymphoma, mantle cell lymphoma, transformed lymphoma, follicular lymphoma (any grade), small lymphocytic lymphoma, marginal zone lymphoma, or Hodgkin lymphoma with at least 2 lines of therapy without a curative treatment options.
6. Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status </= 2.
7. Adequate organ function, as specified below, within 3 weeks before the first dose of study drug: a) Bone marrow reserve consistent with: absolute neutrophil count (ANC) >/=1.5 x 10^9/L; platelet count >/=100 x 10^9/L; hemoglobin >/=9 g/dL without transfusion within 1 week preceding study drug administration; b) Hepatic: total bilirubin < /=1.5 x upper limit of normal (ULN), transaminases (aspartate aminotransferase-AST and alanine aminotransferase ALT) </= 2.5 x ULN (</= 5 x ULN if liver metastases are present); c) Renal: creatinine clearance >/= 50 mL/min based either on Cockcroft-Gault estimate or based on urine collection (12 or 24 hour); d) Metabolic: fasting serum glucose (</=130 mg/dL) and fasting triglycerides </=300 mg/dL;
8. Ability to swallow oral medications;
9. Measurable disease, defined as >/=1.5 cm on imaging assessment.

Exclusion Criteria:

1. Eligible for therapy for the lymphoid malignancy which has a high likelihood of a curative result in the opinion of the investigator.
2. Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening period
3. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
4. Concurrent malignancies except basal or squamous cell carcinoma of the skin, or cervical carcinoma in situ treated with curative intent. Any cancer from which the patient has been disease free for at least 2 years is permissible.
5. Treatment with any investigational products within 14 days before the first dose of study drug
6. Failed to recover to baseline or stable grade 1 from the reversible effects of prior anticancer therapies with the exception of alopecia.
7. Manifestations of malabsorption due to prior gastrointestinal (GI) surgery, GI disease, or for an unknown reason that may alter the absorption of TAK228; such as significant chronic diarrhea. In addition, patients with enteric stomata are also excluded.
8. Poorly controlled diabetes mellitus defined as HbA1c > 7%; subjects with a history of transient glucose intolerance due to corticosteroid administration are allowed in this study if all other inclusion/exclusion criteria are met;
9. History of any of the following within the last 6 months prior to study entry: ischemic myocardial event, including angina requiring therapy and artery revascularization procedures; Ischemic cerebrovascular event, including TIA and artery revascularization procedures; Requirement for inotropic support (excluding digoxin) or serious (uncontrolled) cardiac arrhythmia (including atrial flutter/fibrillation, ventricular fibrillation or ventricular tachycardia); Placement of a pacemaker for control of rhythm; New York Heart Association (NYHA) Class III or IV heart failure; Pulmonary embolism.
10. History of any of the following within the last 6 months prior to study entry: Requirement of inotropic support; Serious uncontrolled cardiac arrhythmia (including atrial flutter/fibrillation, ventricular fibrillation or ventricular tachycardia); Placement of a pacemaker for control of rhythm
11. Significant active cardiovascular or pulmonary disease at the time of study entry, including: uncontrolled high blood pressure (i.e., systolic blood pressure >180 mm Hg, diastolic blood pressure > 95 mm Hg) Use of anti-hypertensive agents to control hypertension before cycle 1 day 1 is allowed; Pulmonary hypertension; Uncontrolled asthma or O2 saturation < 90% by ABG (Arterial Blood Gas) analysis or pulse oximetry on room air; Significant valvular disease; severe regurgitation or stenosis by imaging independent of symptom control with medical intervention, or history of valve replacement; medically significant (symptomatic) bradycardia; History of arrhythmia requiring an implantable cardiac defibrillator; Baseline prolongation of the rate-corrected QT interval (QTc) (e.g., repeated demonstration of QTc interval > 480 milliseconds, or history of congenital long QT syndrome, or torsades de pointes).
12. Treatment with strong inhibitors and/or inducers of cytochrome P450 (CYP) 3A4, CYP2C9 or CYP2C19 within 1 week preceding the first dose of study drug.
13. Patients receiving systemic corticosteroids (either IV or oral steroids, excluding inhalers or low-dose hormone replacement therapy as defined no greater than 20mg of prednisone daily) within 1 week before administration of the first dose of study drug.
14. Other clinically significant co-morbidities, such as uncontrolled pulmonary disease, active central nervous system disease, active infection, or any other condition that could compromise participation of the patient in the study.
15. Central nervous system (CNS) lymphoma.
16. Known human immunodeficiency virus infection.
17. Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection.
18. Diagnosed or treated for another malignancy within 2 years before administration of the first dose of study drug, or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
19. Daily or chronic use of a proton pump inhibitor (PPI) and/or having taken a PPI within 7 days before receiving the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason R. Westin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was open from 03/01/2017 to 11/27/2017
Pre-assignment Details: No significant events in the study occurred after enrollment, prior to assignment to arm/group
Groups:
- Aggressive NHL(DLBCL/MCL/Transformed Large Cell Lymphoma/FL gr: Aggressive NHL(DLBCL/MCL/transformed large cell lymphoma/FL grade 3b
- Indolent NHL:FL grade1-3a,SLL,MZL: Indolent NHL:FL grade1-3a,SLL,MZL
- Hodgkin Lymphoma: Hodgkin lymphoma
Period: Overall Study
Arm/Group | Aggressive NHL(DLBCL/MCL/Transformed Large Cell Lymphoma/FL gr | Indolent NHL:FL grade1-3a,SLL,MZL | Hodgkin Lymphoma
Started | 4 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 4 | 0 | 0
Not completed — Screen Failure | 2 | 0 | 0
Not completed — Progressive disease | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Dr. Westin (Principal Investigator) was only participating in the DLBCL arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aggressive NHL(DLBCL/MCL/Transformed Large Cell Lymphoma/FL gr | Indolent NHL:FL grade1-3a,SLL,MZL | Hodgkin Lymphoma | Total
Number analyzed (Participants) | 4 | 0 | 0 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 3 |  |  | 3
  >=65 years | 1 |  |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  |  | 1
  Male | 3 |  |  | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  |  | 0
  Not Hispanic or Latino | 0 |  |  | 0
  Unknown or Not Reported | 4 |  |  | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 1 |  |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 1 |  |  | 1
  White | 1 |  |  | 1
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 1 |  |  | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 |  |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Response Assessment (RA)
Description: RA was defined by Lugano Criteria & based on CT scans obtained at screening & after completion of every 2 cycles of therapy. Complete Radiographic Response Target Nodes must regress to <=1.5cm in longest dimension,No extralymphatic sites of disease. PR >=50% decrease in sum of the product of diameters of up to 6 target measurable nodes and extranodal sites. When a lesion is too small to measure on CT, 5 mmx5mm is assigned. When not visible on CT, assign 0x0 mm. For a node 5mmx5mm use actual measurement. SD< 50% decrease in sum of the product of diameters of up to 6 target measurable nodes & extranodal sites, no criteria for disease progression are met. Progressive disease requires one of the following:An individual node must be abnormal with: LDi 1.5cm & Increase by 50% from PPD nadir & an increase in LDi or SDi from nadir 0.5cm for lesions 2cm,1cm for lesions 2cm. In case of splenomegaly, the splenic length must increase by >=50% of the extent of its prior increase beyond baseline.
Time Frame: Time frame for response assessment was from Baseline to end of treatment or progression of disease up to 1 year.
Population: No analysis could be performed due to 2 participants failed screening and 2 participants disease progressed before analysis could be performed
Arm/Group | Aggressive NHL(DLBCL/MCL/Transformed Large Cell Lymphoma/FL gr | Indolent NHL:FL grade1-3a,SLL,MZL | Hodgkin Lymphoma
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Progression free survival, duration of response and overall survival analysis could not be properly evaluated due to patients being taken off study early due to progression of disease but safety and tolerability were reported through safety event reports, please see AEs-serious and non-serious section for this.
Time Frame: Baseline to end of treatment or progression of disease
Population: Adverse events were evaluated for the time patients were on study however due to early progression of disease, patients did not finish the treatment and adverse events reported were not conclusive of toxicity related to drug. Updated to two participants for the secondary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Aggressive NHL(DLBCL/MCL/Transformed Large Cell Lymphoma/FL gr | Indolent NHL:FL grade1-3a,SLL,MZL | Hodgkin Lymphoma
Number analyzed (Participants) | 2 | 0 | 0
Participants | 2 |  |

3. Other Pre Specified Outcome: Exploratory Objective to Define Change of mTOR Pathway Protein Phosphorylation and the Incidence of Activating Mutations in MTOR and Related Genes.
Description: Assessed with reverse phase protein arrays after exposure to TAK228,
Time Frame: Baseline to end of treatment or progression of disease
Population: Exploratory objective was not analyzed because patients came off study before it could be analyzed, no data were collected.
Arm/Group | Aggressive NHL(DLBCL/MCL/Transformed Large Cell Lymphoma/FL gr | Indolent NHL:FL grade1-3a,SLL,MZL | Hodgkin Lymphoma
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The time frame for assessment of adverse events was from time of consent to the end of treatment or progression of disease, whichever occurred first.
Description: Adverse events were assessed on 2 patients that were eligible to participate. They were not assessed for 2 patients that were screen failures.
Arm/Group | Aggressive NHL(DLBCL/MCL/Transformed Large Cell Lymphoma/FL gr | Indolent NHL:FL grade1-3a,SLL,MZL | Hodgkin Lymphoma
All-Cause Mortality (participants affected / at risk) | 2/2 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aggressive NHL(DLBCL/MCL/Transformed Large Cell Lymphoma/FL gr (N=2) | Indolent NHL:FL grade1-3a,SLL,MZL (N=0) | Hodgkin Lymphoma (N=0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aggressive NHL(DLBCL/MCL/Transformed Large Cell Lymphoma/FL gr (N=2) | Indolent NHL:FL grade1-3a,SLL,MZL (N=0) | Hodgkin Lymphoma (N=0)
Edema Limbs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Renal insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Anorexia/appetite change (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (right thigh) (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | NA
Diarrhea (Gastrointestinal disorders) | 1 (1) | NA | NA
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | NA | NA
Blurred vision (Eye disorders) | 1 (1) | NA | NA
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT02727777/Prot_SAP_000.pdf